CLINICAL TRIAL: NCT04744298
Title: Identification and Treatment of Hypoxemic Respiratory Failure (HRF) and ARDS With Protection, Paralysis, and Proning: TheraPPP Study
Brief Title: Identification and Treatment of Hypoxemic Respiratory Failure and ARDS With Protection, Paralysis, and Proning Pathway
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Principal Investigator, Ken Kuljit Parhar, MD, Consultant Intensivist & Clinical Assistant Professor Affiliation: University of Calgary, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB20-0646
Record Dates: First submitted 2021-02-01; First posted 2021-02-08 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Acute Respiratory Distress Syndrome; Hypoxemic Respiratory Failure; ARDS, Human
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: The study uses an effectiveness-implementation hybrid design (type 1). Phase 1 will evaluate effectiveness and Phase 2 will assess the implementation of the pathway. Implementation will occur via a pragmatic registry-based stepped wedge cluster randomization of ICUs. The unit of randomization will be a cluster of 2 ICUs. The intervention will be implemented into 1 cluster every 2 months. Once implemented, the cluster will continue to receive it for the remainder of the study.
  Effectiveness: There will be a 10-month baseline data collection period at the beginning of the study. The total study duration will be 29 months (Estimated18816 mechanically ventilated patients including 2688 in the ARDS subgroup). The comparison (control) therapy will be usual management assessed in the baseline period.
  Implementation: A process evaluation of pathway implementation will be conducted to 1) quantitatively evaluate fidelity, 2) qualitatively assess acceptability (Estimate 1100 clinicians).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TheraPPP Pathway (Experimental): The investigators will perform an effectiveness-implementation hybrid study design (type 1) to evaluate the effectiveness and implementation of the TheraPPP pathway.
  All mechanically ventilated patients admitted to the ICU will enter the pathway. To evaluate effectiveness the investigators will collect patient data for approximately 29 months. To assess acceptability of the pathway the investigators will conduct a survey and focus groups to clinicians who used the Pathway.
  Interventions: Other: TheraPPP

INTERVENTIONS:
Other: TheraPPP — TheraPPP Steps:
  Step 1. All mechanically ventilated patients will have a height measured and documented. Step 2. Screening for HRF. Step 3. Initiate Lung Protective Ventilation (LPV). Step 4. Paralysis. Step 5. Prone Positioning.

SUMMARY:
Treatment of patients with Hypoxemic respiratory failure (HRF) and Acute Respiratory Distress Syndrome (ARDS) is complex. Therapies that have been shown to save the lives of patients with HRF and ARDS are available but they are not always provided. To reduce practice variation and improve adherence to evidence-informed therapies, the investigators developed the Treatment of Hypoxemic Respiratory Failure and ARDS with Protection, Paralysis, and Proning (TheraPPP) Pathway.

The overall objective of TheraPPP Pathway is to improve the quality of care for patients with HRF. Implementation of the pathway across Alberta will test the effectiveness and implementation of the TheraPPP Pathway.

DETAILED DESCRIPTION:
Hypoxemic respiratory failure (HRF) and ARDS are common conditions among patients admitted to the Intensive care unit (ICU). Treatment of these patients is complex. Evidence based therapies that can improve survival exist; however, implementation is extremely inconsistent. As a potential solution to this problem, the investigators developed the Treatment of Hypoxemic Respiratory Failure (HRF) and ARDS with Protection, Paralysis, and Proning (TheraPPP) Pathway to reduce practice variation and improve adherence to evidence-informed therapy.

The TheraPPP pathway is a comprehensive evidence-based, stakeholder-informed pathway for the diagnosis and management of HRF. The overall objective of the pathway is to improve the quality of care for patients with HRF. The specific objectives are to evaluate:

1. Effectiveness of the pathway. A cost-effectiveness analysis is a secondary objective.
2. Implementation of the pathway by conducting a process evaluation which will assess fidelity of the delivered interventions and clinician perceptions about the acceptability of the pathway.

Mechanically ventilated patients admitted to any one of 17 adult ICUs in Alberta will receive the intervention. One ICU (Calgary) is the setting for a pilot study (NCT04070053).

For data analysis, the investigators will use chart abstraction to quantitatively assess the fidelity of the delivered intervention, and surveys and focus groups to qualitatively assess clinician perceptions about the acceptability of the pathway. Fidelity of the intervention will be tracked using process of care indicators that reflect the five key steps of the pathway.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the one of the 17 adult Intensive Care Units in Alberta
* Invasively mechanically ventilated

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19916 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
EFFECTIVENESS (primary clinical outcome) 28-day ventilator free days | 4 months (after the study post-intervention period)
  A composite outcome of survival and days spent not ventilated over the first 28 days
IMPLEMENTATION (primary fidelity outcome) Composite Fidelity Score | 4 months (after the study post-intervention period)
  The composite fidelity score is measured daily for each patient. It is scored out of 5 and awards 1 point for each fidelity indicator (listed below) that investigators are able to measure:
  1. If ventilated, is a height measured (step 1)
  2. If arterial to inspired oxygen ratio (PaO2:FiO2 ratio or PF ratio) ≤300, is the medial tidal volume ≤8mL/kg (step 2)
  3. If PF ratio ≤300, is a plateau pressure measured (step 3)
  4. IF patient has HRF and PF ratio ≤150, was neuromuscular blockade used in that 24 hour period (step 4)
  5. If the patient has HRF and PF ratio ≤150 and FiO2 ≥0.6, did the patient receive prone ventilation (step 5)
ECONOMIC (primary economic outcome) Cost per ventilator free day saved | 4 months (after the study post-intervention period)
  Cost per ventilator free day saved from the perspective of the health care system over the index hospitalization period

SECONDARY OUTCOMES:
28-day and hospital survival | 90 days
  Number of patients who die in the ICU, hospital, and at or before 28-day hospital censored at 90 days
Ventilator duration | 4 months (after the study post-intervention period)
  The number of ventilated days. If a patient is invasively mechanically ventilated via endotracheal tube or tracheostomy for any period of time in a 24 hour period (0000-2359) this is considered a ventilated day. A ventilated day is the component of VFDs that reflects duration of ventilation.
Driving Pressure | 4 months (after the study post-intervention period)
  Calculated on patients ventilated with PF ratio (partial pressures of oxygen (paO2) / fraction of inspired oxygen (FiO2) ≤ 300 on a controlled mode as plateau pressure - positive end expiratory pressure (PEEP).
Mechanical Power | 4 months (after the study post-intervention period)
  Calculated on patients ventilated with PF ratio ≤ 300 on a controlled mode using the formula Power = 0.098*respiratory rate•(tidal volume/1000)*(Peak Pressure - (0.5 • Driving Pressure)).
ICU and hospital length of stay | 4 months (after the study post-intervention period)
  The number of days that patients stay in the ICU and in hospital
Proportion of patients receiving rescue therapies specifically Extracorporeal Life Support (ECLS) | 4 months (after the study post-intervention period)
  The proportion of patients receiving rescue therapies including ECLS
The proportion of patients ventilated with a height measured | 4 months (after the study post-intervention period)
  Total number of ventilated patients for with a height measured divided by the total number of patients ventilated
Proportion of patient days with PF ratio ≤300 with a tidal volume ≤8mL/kg | 4 months (after the study post-intervention period)
  The total number of patient days with arterial to inspired oxygen ratio(PaO2:FiO2 ratio or PF ratio) ≤300 with a tidal volume ≤8 mL/kg divided by the total number of of patient days with arterial to inspired oxygen ratio (PaO2:FiO2 ratio or PF ratio) ≤300
Proportion of patient days with PF ratio ≤300 with a plateau pressure measured | 4 months (after the study post-intervention period)
  The total number of patient days with PF ratio ≤300 with a plateau pressure measured divided by the total number of patient days with PF ratio ≤300
Proportion of patient days with HRF and PF ratio ≤150 who receive neuromuscular blockade | 4 months (after the study post-intervention period)
  The number of patient days with HRF and PF ratio ≤150 who receive neuromuscular blockade divided by the number of patient days with HRF and PF ratio ≤150
Proportion of patient days with HRF and PF ratio ≤150 and FiO2 ≥0.6 receiving prone ventilation | 4 months (after the study post-intervention period)
  The number of patient days with HRF and PF ratio ≤150 and FiO2 ≥0.6 receiving prone ventilation divided by the number of patient days with HRF and PF ratio ≤150 and FiO2 ≥0.6
Theoretical Framework of Acceptability - Composite Acceptability Score | 4 months (after the study post-intervention period)
  Pathway acceptability is measured using the Theoretical Framework of Acceptability (TFA). The primary outcome for acceptability is a composite score of the proportion of seven TFA constructs [(1) affective attitude (2) burden (3) ethicality (4) intervention coherence (5) opportunity costs (6) perceived effectiveness (7) self-efficacy] graded with a median score of 4 or above from a 5-point Likert scale, in which 1 indicates strong disagreement (and lower acceptability) and 5 indicates strong agreement (and higher acceptability).
Theoretical Framework of Acceptability - Opportunity costs construct | 4 months (after the study post-intervention period)
  Benefits or costs to the participant for using the pathway graded on a 5-point Likert scale in which 1 indicates strong disagreement (and lower acceptability) and 5 indicates strong agreement (and higher acceptability), Median (IQR)
Theoretical Framework of Acceptability - Perceived effectiveness construct | 4 months (after the study post-intervention period)
  The extent to which the intervention is perceived as likely to achieve its purpose graded graded on a 5-point Likert scale in which 1 indicates strong disagreement (and lower acceptability) and 5 indicates strong agreement (and higher acceptability), Median (IQR)
Theoretical Framework of Acceptability - Affective attitude construct | 4 months (after the study post-intervention period)
  How an individual feels about the intervention graded on a 5-point Likert scale in which 1 indicates strong disagreement (and lower acceptability) and 5 indicates strong agreement (and higher acceptability), Median (IQR)
Theoretical Framework of Acceptability - Burden construct | 4 months (after the study post-intervention period)
  The perceived amount of effort that is required to participate in the intervention graded on a 5-point Likert scale in which 1 indicates strong disagreement (and lower acceptability) and 5 indicates strong agreement (and higher acceptability), Median (IQR)
Theoretical Framework of Acceptability - Ethicality construct | 4 months (after the study post-intervention period)
  The extent to which the intervention has a good fit with an individual's value graded on a 5-point Likert scale in which 1 indicates strong disagreement (and lower acceptability) and 5 indicates strong agreement (and higher acceptability), Median (IQR)
Theoretical Framework of Acceptability - Self efficacy construct | 4 months (after the study post-intervention period)
  The participant's confidence that they can perform the behavior(s) required to participate in the intervention graded on a 5-point Likert scale in which 1 indicates strong disagreement (and lower acceptability) and 5 indicates strong agreement (and higher acceptability), Median (IQR)
Theoretical Framework of Acceptability - Intervention coherence construct | 4 months (after the study post-intervention period)
  The extent to which the participant understands the invention and how it works graded on a 5-point Likert scale in which 1 indicates strong disagreement (and lower acceptability) and indicates strong agreement (and higher acceptability), Median (IQR)
Total cost: ICU admission | 4 months (after the study post-intervention period)
  Total cost for the ICU admission
Total cost: Index hospitalization | 4 months (after the study post-intervention period)
  Total cost for the index hospitalization
Cost per quality adjusted life year (QALY) | 4 months (after the study post-intervention period)
  Cost per quality adjusted life year (QALY) from the health care system perspective over the patient's lifetime

CONTACTS AND LOCATIONS:
Overall Officials: Ken K Parhar, MD, MSc, Principal Investigator — University of Calgary
Locations (17):
- Canada (17):
  - Peter Lougheed Centre (PLC), Calgary, Alberta
  - Foothills Hospital Intensive Care Unit, Calgary, Alberta
  - Foothills Medical Center Cardiovascular ICU, Calgary, Alberta
  - Rockyview General Hospital, Calgary, Alberta
  - South Health Campus, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Misericordia Community Hospital, Edmonton, Alberta
  - Mazankowski Alberta Heart Institute, Edmonton, Alberta
  - University of Alberta Hospital General Systems ICU, Edmonton, Alberta
  - University of Alberta Hospital Neurosciences Intensive Care Unit, Edmonton, Alberta
  - Grey Nuns Community Hospital, Edmonton, Alberta
  - Northern Lights Regional Health Centre, Fort McMurray, Alberta
  - Queen Elizabeth II Hospital, Grande Prairie, Alberta
  - Chinook Regional Hospital, Lethbridge, Alberta
  - Medicine Hat Regional Hospital, Medicine Hat, Alberta
  - Red Deer Regional Hospital Centre, Red Deer, Alberta
  - Sturgeon Community Hospital, St. Albert, Alberta

REFERENCES:
- [Derived] Krewulak KD, Knight G, Irwin A, Morrissey J, Stelfox HT, Bagshaw SM, Zuege D, Roze des Ordons A, Fiest K, Parhar KKS. Acceptability of the Venting Wisely pathway for use in critically ill adults with hypoxaemic respiratory failure and acute respiratory distress syndrome (ARDS): a qualitative study protocol. BMJ Open. 2024 May 28;14(5):e075086. doi: 10.1136/bmjopen-2023-075086. PMID 38806421
- [Derived] Parhar KKS, Soo A, Knight G, Fiest K, Niven DJ, Rubenfeld G, Scales D, Stelfox HT, Zuege DJ, Bagshaw S. Protocol and statistical analysis plan for the identification and treatment of hypoxemic respiratory failure and acute respiratory distress syndrome with protection, paralysis, and proning: A type-1 hybrid stepped-wedge cluster randomised effectiveness-implementation study. Crit Care Resusc. 2023 Dec 13;25(4):207-215. doi: 10.1016/j.ccrj.2023.10.008. eCollection 2023 Dec. PMID 38234326

DOCUMENTS (2):
  • Study Protocol (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/98/NCT04744298/Prot_002.pdf
  • Statistical Analysis Plan (2022-02-22): https://cdn.clinicaltrials.gov/large-docs/98/NCT04744298/SAP_001.pdf